CLINICAL TRIAL: NCT02746068
Title: COAST -1: Clinical Knee Osteoarthritis Symptom Treatment 1 Study. A Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of AXS-02 (Disodium Zoledronate Tetrahydrate) Administered Orally to Subjects With Knee Osteoarthritis Associated With Bone Marrow Lesions.
Brief Title: A Study to Assess the Efficacy and Safety of AXS-02 in Subjects With Knee OA Associated With Bone Marrow Lesions
Acronym: COAST-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXS02-K301
Record Dates: First submitted 2016-04-14; First posted 2016-04-21 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Bone Marrow Lesions; AXS02; Axsome; Knee OA; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AXS-02 (Experimental): Administered orally in the morning for 6 weeks
  Interventions: Drug: AXS-02
- Placebo (Placebo Comparator): Administered orally in the morning for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-02
  Arms: AXS-02
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 24-week study to evaluate the efficacy and safety of AXS-02 in subjects with knee osteoarthritis associated with bone marrow lesions.

ELIGIBILITY:
Key Inclusion Criteria:

* Male at least 50 years of age, or postmenopausal female
* Meets the ACR clinical criteria for knee osteoarthritis
* Bone Marrow Lesion of the knee present on MRI
* Additional criteria may apply

Key Exclusion Criteria:

* Previous surgery on index knee
* Any prior use of bisphosphonates within 6 months of screening
* Additional criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported pain intensity | Baseline to Week 24
  Patient reported pain intensity is recorded as an average daily pain intensity using an 11-point scale (0 = no pain to 10 = worst pain possible)

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGI-C) | Week 12 and Week 24
Clinical Global Impression of Change (CGI-C) scores | Week 12 and Week 24
Change in WOMAC pain and stiffness subscales over time | Baseline to Week 24

CONTACTS AND LOCATIONS:
Locations (61):
- United States (54):
  - Achieve Clinical Research, Birmingham, Alabama
  - Birmingham, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Hot Springs, Arkansas
  - Anaheim, California
  - Canoga Park, California
  - El Cajon, California
  - La Mesa, California
  - Long Beach, California
  - Los Angeles, California
  - North Hollywood, California
  - Sacramento, California
  - San Diego, California
  - Thousand Oaks, California
  - Upland, California
  - Denver, Colorado
  - Milford, Connecticut
  - Boynton Beach, Florida
  - Clearwater, Florida
  - Clermont, Florida
  - Hialeah, Florida
  - Jupiter, Florida
  - Lauderdale Lakes, Florida
  - Orlando, Florida
  - Accord Clinical Research, Port Orange, Florida
  - Port Saint Lucie, Florida
  - Sarasota, Florida
  - Canton, Georgia
  - Chicago, Illinois
  - Affinity Clinical Research Institute, Oak Lawn, Illinois
  - Oak Lawn, Illinois
  - Newton, Kansas
  - Wheaton, Maryland
  - Boston, Massachusetts
  - North Attleboro, Massachusetts
  - Quincy, Massachusetts
  - Kansas City, Missouri
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Hartsdale, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Duncansville, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Franklin, Tennessee
  - Austin, Texas
  - Baytown, Texas
  - DeSoto, Texas
  - Wichita Falls, Texas
  - Newport News, Virginia
  - Bellevue, Washington
- Australia (7):
  - Broadmeadow, New South Wales
  - Noosa, Queensland
  - Adelaide, South Australia
  - Hobart, Tasmania
  - Clayton, Victoria
  - Melbourne, Victoria
  - Nedlands, Western Australia